CLINICAL TRIAL: NCT03444454
Title: The Italian Network of Telerehabilitation: Evaluation of Telerehabilitation System for Continuum of Care in Multiple Sclerosis
Brief Title: Telerehabilitation in Multiple Sclerosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: IRCCS Centro Neurolesi Bonino Pulejo (Other); Fondazione Mondino (Other); IRCCS San Camillo, Venezia, Italy (Other); IRCCS San Raffaele Roma (Other); Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Principal Investigator, Francesca Baglio, MD, researcher, Fondazione Don Carlo Gnocchi Onlus
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FdG_VRRS_MS_01
Record Dates: First submitted 2018-02-02; First posted 2018-02-23 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis
Keywords: Telerehabilitation; Virtual reality; Quality of life; transcranial Direct Current Stimulation
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- VRRS Khymeia (Experimental): The group will receive a kit home-based (a tablet home, an exercise equipment, access to a daily individualized training program).
  The exercise program will be remotely charged by therapist on the patient's computer.
  Each patient's performed session will be reviewed remotely by the therapist.
  Interventions: Behavioral: VRRS Khymeia
- Usual care program (Active Comparator): The usual care group will have written, home-based exercise program, provided to them at an initial face-to-face assessment.
  Interventions: Behavioral: Usual care program
- VRRS Khymeia plus active tDCS (Experimental): The group will receive 5 sessions each lasting 45 minutes of an individualized home-based VRRS training combined with active (anodal) tDCS applied to the left dorsolateral prefrontal cortex over 1 week, followed by 5 weeks of home-based VRRS training
  Interventions: Behavioral: VRRS Khymeia plus active tDCS
- VRRS Khymeia plus placebo tDCS (Active Comparator): The group will receive 5 sessions of an individualized home-based VRRS training combined with placebo tDCS applied to the left dorsolateral prefrontal cortex over 1 week, followed by 5 weeks of home-based VRRS training
  Interventions: Behavioral: VRRS Khymeia plus placebo tDCS

INTERVENTIONS:
Behavioral: VRRS Khymeia — Participants will receive an individualized exercise program set up by the therapist. The intervention applied to the experimental group will consist of 30 sessions of Khymeia VRRS training distributed in five sessions for week, each lasting 45 minutes.
  Each session is constructed by alternating physical with cognitive activities. The sessions will initially be tailored to the patient's baseline characteristics. Remotely, the therapist will then adjust the participant's exercise program as appropriate, by changing exercises, level of difficulty or number of repetitions.
  Arms: VRRS Khymeia
Behavioral: Usual care program — The usual care group will have written, home-based exercise program, provided to them at an initial face-to-face assessment.
  Arms: Usual care program
Behavioral: VRRS Khymeia plus active tDCS — Participants will receive 5 sessions each lasting 45 minutes of an individualized home-based VRRS training combined with active (anodal) tDCS applied to the left dorsolateral prefrontal cortex over 1 week, followed by 5 weeks of home-based VRRS training.
  The sessions of VRRS will initially be tailored to the patient's baseline characteristics. Remotely, the therapist will then adjust the participant's exercise program as appropriate, by changing exercises, level of difficulty or number of repetitions.
  Arms: VRRS Khymeia plus active tDCS
Behavioral: VRRS Khymeia plus placebo tDCS — Participants will receive 5 sessions each lasting 45 minutes of an individualized home-based VRRS training combined with active (anodal) tDCS applied to the left dorsolateral prefrontal cortex over 1 week, followed by 5 weeks of home-based VRRS training.
  The sessions of VRRS will initially be tailored to the patient's baseline characteristics. Remotely, the therapist will then adjust the participant's exercise program as appropriate, by changing exercises, level of difficulty or number of repetitions.
  Arms: VRRS Khymeia plus placebo tDCS

SUMMARY:
The main aim of the study is to evaluate the efficacy of the Virtual Reality Rehabilitation System (VRRS, Khymeia) compared to usual care treatment for patients with MS at home.

The effects of the intervention on outcome variables will be assessed using a randomized controlled trial design with a comparison group receiving usual care training. The investigators will assess the effect of VRRS system on the quality of life, motor, and cognitive abilities. (Phase I) In the second phase of the present study we aim to evaluate the effects induced by the treatment of active (anodal) transcranial Direct Current Stimulation (tDCS) applied to the left dorsolateral prefrontal cortex (lDLPFC) combined with VRRS compared to placebo tDCS stimulation combined with VRRS. The effects of the intervention patient-relevant outcomes will be assessed using a randomized controlled trial design with four groups. The investigators will assess the effect of VRRS system on patient-relevant outcomes motor, cognitive and participation. (Phase II)

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Multiple Sclerosis (RR and SP) based on McDonald criteria
* Education ≥ 8 ages
* Italian mother language
* Right-handedness
* Use of corticosteroids for three months prior to the study, having and no acute exacerbations of symptoms within three months of the study.

Exclusion Criteria:

* Existence of visual acuity and acoustic perception problems, to prevent performance of VRRS activities
* Relapses next to the time of enrolment (3 months)
* EDSS > 6.5.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in measure of quality of life | Baseline up to 6 weeks and 6 months
  Quality of life will be measured by 54-item Multiple Sclerosis Quality of Life (MSQOL-54) questionnaire
  There is no single overall score for the MSQOL-54. Two summary scores - physical health and mental health - can be derived from a weighted combination of scale scores. In addition, there are 12 subscales: physical function, role limitations-physical, role limitations-emotional, pain, emotional well-being, energy, health perceptions, social function, cognitive function, health distress, overall quality of life, and sexual function. There are also two single-item measures: satisfaction with sexual function and change in health.
  Administration forms and scoring instructions can be downloaded (https://www.nationalmssociety.org/NationalMSSociety/media/MSNationalFiles/Brochures/MSQOL54_995.pdf ).
  Higher values represent a better outcome

SECONDARY OUTCOMES:
Change in balance | Baseline up to 6 weeks and 6 months
  Mini-Balance Evalutation System (mini-BES) Test
Change in gait | Baseline up to 6 weeks and 6 months
  12-item Multiple Sclerosis Walking Scale
Change gross manual dexterity | Baseline up to 6 weeks and 6 months
  Box and Block Test
Change in global cognitive status | Baseline up to 6 weeks and 6 months
  Montreal Cognitive Assessment (MoCA) test
Change cognitive status | Baseline up to 6 weeks and 6 months
  Symbol Digit Modalities Test (Form Brief Repeatable Battery of Neuropsychological Tests )
Change in fatigue | Baseline up to 6 weeks and 6 months
  Fatigue Severity Scale
  A questionnaire with 9 items (questions)
  Grading of each FSS item ranges from 1 to 7, where 1 indicates strong disagreement and 7 strong agreement, and the final score represents the mean value of the 9 items
  Higher values represent a worse outcome
Change in Emotional Traits | Baseline up to 6 weeks and 6 months
  The Regulatory Emotional Self-Efficacy (RESE) scale
  The RESE scale assesses self-efficacy in expressing positive emotions and self-efficacy in managing negative emotions.
  With this scale, participants rate (ranging from 1 [not well at all] to 5 [very well]) their capability to manage their emotional life. RESE scale consists of 12 items and are calculated 3 scores: 1) self-efficacy in expressing positive emotions (POS) score; 2)self-efficacy in managing negative emotions (NEG) score; 3)self-efficacy in managing despondency/distress (DES) score
  Higher values within each score represent a better outcome
Change in Behavioral (depression) | Baseline up to 6 weeks and 6 months
  Beck Depression Inventory
Change in Behavioral (anxiety) | Baseline up to 6 weeks and 6 months
  State-trait anxiety inventory

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Fondazione Don Carlo Gnocchi, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Di Tella S, Pagliari C, Blasi V, Mendozzi L, Rovaris M, Baglio F. Integrated telerehabilitation approach in multiple sclerosis: A systematic review and meta-analysis. J Telemed Telecare. 2020 Aug-Sep;26(7-8):385-399. doi: 10.1177/1357633X19850381. Epub 2019 May 27. PMID 31132909
- [Derived] Pagliari C, Di Tella S, Jonsdottir J, Mendozzi L, Rovaris M, De Icco R, Milanesi T, Federico S, Agostini M, Goffredo M, Pellicciari L, Franceschini M, Cimino V, Bramanti P, Baglio F. Effects of home-based virtual reality telerehabilitation system in people with multiple sclerosis: A randomized controlled trial. J Telemed Telecare. 2024 Feb;30(2):344-355. doi: 10.1177/1357633X211054839. Epub 2021 Dec 1. PMID 34851211